CLINICAL TRIAL: NCT04380922
Title: Prevalence of Periodontal Diseases in Inflammatory Bowel Diseases : a Pilot-study
Brief Title: Prevalence of Periodontal Diseases in IBD
Acronym: MICIMaP
Status: Completed | Type: Observational
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Other Study IDs: PO20062*
Record Dates: First submitted 2020-05-05; First posted 2020-05-08 (Actual); Last update posted 2022-06-13 (Actual); Status verified 2022-06

CONDITIONS: Inflammatory Bowel Diseases; Periodontal Diseases
MeSH Terms: conditions — Inflammatory Bowel Diseases; Periodontal Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Active IBD: Active Inflammatory Bowel Diseases defined as :
  For Crohn's disease :
  * Harvey Bradshaw Index ≥ 4
  * Associated with fecal calprotectin rate > 250 µg/g within 3 months OR CRP ≥ 6mg /L OR the presence of ulcerative and/or inflammatory lesions in endoscopy or in imaging within 3 months For Ulcerative colitis
  * Partial Mayo score ≥ 2
  * Associated with fecal calprotectin rate > 250 µg/g within 3 months OR CRP ≥ 6mg /L OR the presence of ulcerative and/or inflammatory lesions in endoscopy within 3 months
  Interventions: Other: Periodontal screening
- Non-active IBD: Non-active Inflammatory Bowel Diseases
  Interventions: Other: Periodontal screening

INTERVENTIONS:
Other: Periodontal screening — Periodontal data collection (PPD, REC, CAL)

SUMMARY:
Periodontal diseases are highly prevalent inflammatory diseases. It is now well known that they are correlated with numerous systemic diseases as : diabetes, chronic obstructive pulmonary disease, metabolic syndrome or rheumatoid arthritis. Recently, periodontal diseases have been correlated with inflammatory bowel diseases (IBD). IBD include two types, Crohn's disease and Ulcerative Colitis. It could be a significant risk factor for the pathogenesis of periodontal disease. These diseases present common features : a high prevalence worldwide, multifactorial pathogenies with common mechanisms. To date, no study has linked activity of IBD and periodontal diseases. The authors hypotheses that the prevalence of periodontal diseases could be increased in patient presenting an active IBD

DETAILED DESCRIPTION:
The present study explores the prevalence of periodontal diseases regarding to the activity status of IBD (active versus non-active).

Diseases activity will be assessed by HBI (Crohn's disease) or partial Mayo score (Ulcerative Colitis) associated with fecal calprotectin and/or CRP and/or inflammatory/ulcerative lesions.

Periodontal diseases (periodontitis and gingivitis) will be diagnosed according to the international classification of periodontal diseases (Chicago 2017) and based on the decision-making algorithms by Tonetti and Sanz. A periodontal screening, socio-demographic data and clinical data will be collected. Then, oral mucosa dermatological manifestations relative to IBD, treatment need (ICDAS) and quality of life related to oral health (GOHAI) will be evaluated. These data will be collected by a periodontist.

The principal hypothesis of this study is that the prevalence of periodontal diseases could be increased in patient presenting an active IBD.

The primary objective is to evaluate if patients presenting active IBD present more stage III and IV periodontal diseases than non-active IBD ones.

The second objectives are :

* to compare periodontal diseases, gingivitis and oral mucosa dermatological manifestations rates according to the diseases activity, the IBD type and the treatment used to treat IBD,
* to compare oral treatment need according to the activity and the type of IBD,
* to compare quality of life related to oral health according to the activity and the type of IBD

ELIGIBILITY:
Inclusion Criteria:

Patients

* consulting Gastroenterology departments in the university hospital of Reims or Amiens-Picardie for the management of Crohn's disease or Ulcerative colitis
* signed informed consent form
* affiliated to the French Social Security system

Exclusion Criteria:

Patients presenting:

* a medical history likely to compromise protocol (psychiatric disorders, other inflammatory diseases, antibiotics, NSAIDs within the last 3 months)
* Diabetes
* Inflammatory rheumatism
* Cancer or radiotherapy up to5 years before inclusion
* X-ray therapy in the area of interest
* Pregnancy or Breastfeeding
* Eating disorders
* Patients under legal protection, trusteeship or guardianship

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients consulting for the management of Crohn's disease or Ulcerative colitis
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2020-06-19 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2022-06-10 (Actual)

PRIMARY OUTCOMES:
Prevalence of Periodontal Disease | Day 0
  Periodontal Disease will be diagnosed according to the new classification of periodontal diseases (Chicago, 2017) and defined by the decision-making algorithms (Tonetti and Sanz, 2019). Diagnosis will be based on Buccal or lingual Clinical attachment level (CAL), Recession (REC) and Periodontal Pocket Depths (PPD) measurement.

SECONDARY OUTCOMES:
Gingivitis | Day 0
  Gingivitis will be diagnosed according to the new classification of periodontal diseases (Chicago, 2017) and defined by the decision-making algorithms (Tonetti and Sanz, 2019). Bleeding On Probing (BOP) higher than 10% is considered as a Gingivitis
Oral mucosa dermatological manifestations secondary to IBD | Day 0
  Defined by WHO criteria (2013)
Oral Health Quality of Life | Day 0
  GOHAI validated in French for general population -Tubert-Jeanin et al., 2003)
Oral treatment need | Day 0
  Evaluated by ICDAS (International Caries Detection and Assessment Score) (Ismaïl et al., 2007)

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Reims, Reims, France

IPD SHARING:
Plan to Share IPD: Undecided